CLINICAL TRIAL: NCT05890612
Title: Post Marketing Surveillance to Observe Safety and Effectiveness of PAXLOVID in Patients With Positive Results of Viral Testing, and Who Are at High Risk for Progression to Severe COVID-19
Brief Title: A Study on Paxlovid Once in the Market, to Observe Its Safety and Effectiveness in Patients Who Have a High Chance of Getting Severe COVID-19
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671020; NCT05890612 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-06-02; First posted 2023-06-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); PAXLOVID; post marketing surveillance (PMS); Korea
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants receiving PAXLOVID: Participants receiving PAXLOVID according to locally approved label.

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of PAXLOVID in the real world and not in clinical studies. The study observes patients who have a high chance of getting severe COVID-19 in Korea.

This study is seeking participants who are:

* Patients with mild-to-moderate COVID-19 symptoms and at high chance of getting severe COVID-19, including hospitalization or death.
* Patients who received, are currently receiving, or are going to receive PAXLOVID according to locally approved label.
* Patients who have signed informed consent documents after understanding all the important parts of the study.

All participants are treated according to routine medical practice and there are no scheduled visits required by this study. All participants will be studied for a follow-up period of 28 days from the last PAXLOVID treatment to understand the safety and the effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received, are currently receiving, or are going to receive PAXLOVID according to locally approved label.
* Patients (or a legally acceptable representative) who are willing to provide written informed consent/assent prior to study enrollment.

Exclusion Criteria:

* Patients with contraindication according to locally approved label of PAXLOVID.
* Patients who are going to receive any investigational medicine during the observation period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received, are currently receiving, or are going to receive PAXLOVID according to locally approved label.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2029-07-13 (Estimated); Study Completion 2029-07-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an adverse event (AE) | Baseline through Day 33
  The number of AEs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with an adverse drug reaction (ADR) | Baseline through Day 33
  The number of ADRs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with a serious AE (SAE) | Baseline through Day 33
  The number of SAEs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with a serious ADR (SADR) | Baseline through Day 33
  The number of SADRs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with an unexpected AE (UAE) | Baseline through Day 33
  The number of UAEs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with an unexpected ADR (UADR) | Baseline through Day 33
  The number of UADRs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with a serious unexpected AE (SUAE) | Baseline through Day 33
  The number of SUAEs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of patients with a serious unexpected ADR (SUADR) | Baseline through Day 33
  The number of SUADRs experienced, the incidence rate, and the number of occurrences among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of COVID-19-related hospitalization from any cause | Baseline through Day 33
  The number and rate of COVID-19-related hospitalizations among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of COVID-19-related death from any cause | Baseline through Day 33
  The number and rate of COVID-19-related deaths among all subjects who received the drug and received at least one safety evaluation will be measured.
Proportion of subjective assessment of COVID-19-related symptomatic change | Day 5, Day 14, Day 33
  The rate of subjective assessment change (improve/no change/worsened) compared to the baseline for COVID-19-related overall symptoms of all subjects who received the drug and received at least one safety evaluation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671020